CLINICAL TRIAL: NCT02255084
Title: Attitude of Unscreened Women Face to Different Strategies to Participate in Cervical Cancer Screening by Vaginal Self-sampling : Home-mailed or Invitation to Remove to Their General Practitioner
Brief Title: Vaginal Self-sampling and Human Papillomavirus Testing in Unscreened Women
Acronym: APACHE-3
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Tours (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Screening
Other Study IDs: INCA13-KH / APACHE-3
Record Dates: First submitted 2014-09-29; First posted 2014-10-02 (Estimated); Last update posted 2025-12-22 (Actual); Status verified 2025-12

CONDITIONS: Cancer Cervix
Keywords: Cervical cancer screening; High Risk Human papillomavirus Infection; vaginal self-sampling; pap smear; general practitioner
MeSH Terms: conditions — Uterine Cervical Neoplasms | interventions — Papanicolaou Test

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Group 1 (Experimental): Group 1 remove self sample kit at gp consulting room or perform pap smear :
  Study coordinators send mail inviting women to remove a kit for vaginal self-sampling at their general practitioner s consulting room.
  Either a pap smear is perform or, at home, women perform vaginal self sampling. Then women send it to a central laboratory for HPV test (Human papillomaVirus).
  Interventions: Behavioral: Group 1 remove self sample kit at gp consulting room or perform pap smear
- Group 2 (Experimental): Group 2 perform self sample at home or pap smear :
  Kit for vaginal self-sampling sent at women home. Women perform vaginal self sampling. Then women send it to a central laboratory for HPV test (Human papillomaVirus).
  Interventions: Behavioral: Group 2 perform self sample at home or pap smear

INTERVENTIONS:
Behavioral: Group 1 remove self sample kit at gp consulting room or perform pap smear — Selected general practitioners are briefly informed about the study and they receive a package of kits for vaginal self-sampling.
  Selected women receive a mail inviting them either to remove a kit for vaginal self-sampling at their general practitioner's consulting room or to perform a pap smear. When women choose the vaginal self-sampling, a HPV test is performed on the sample in a virology laboratory.
  Arms: Group 1
Behavioral: Group 2 perform self sample at home or pap smear — Selected general practitioners are briefly informed about the study. Selected women receive a mail inviting them either to perform a vaginal self sampling at their home (with the kit provided) or to perform a pap smear.
  When women choose the vaginal self-sampling, a HPV test is performed on the sample in a virology laboratory.
  Arms: Group 2

SUMMARY:
Despite the existence of an effective screening test (pap smear), cervical cancer is, every year in France, the cause of more than 3,000 new cases and 1,100 deaths. But, in France, 4 in 10 women are not screened or not often enough (nearly 7 millions women). It is therefore necessary to develop new strategies to reach these women. The etiological factor of this cancer is persistent infection with High-Risk Human PapillomaVirus oncogene (HR-HPV). Thereby, HPV-based tests could be alternative screening tests. Vaginal self-sampling with HR-HPV test is simpler and less intrusive than the pap smear. It has been shown that vaginal self-sampling with HPV test is a powerful means to increase the participation rate in cervical cancer screening.

ELIGIBILITY:
Inclusion Criteria:

* women from 30 to 65 years old
* women living in french territorial division 37 ("Indre-et-Loire")
* women having a reported general practitioner in french territorial division 37 ("Indre-et-Loire")

Exclusion Criteria:

* pap smear made in the three last years

Ages: 30 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3612 (Actual)
Dates: Start 2015-02; Primary Completion 2016-09 (Actual); Study Completion 2016-09 (Actual)

PRIMARY OUTCOMES:
Participation / no participation to complete cervical cancer screening | 9 months after postal mail
  Uncompleted cervical cancer screening is defined as one of the followings :
  * no pap smear
  * no vaginal self-sampling
  * noninterpretable HPV test result and no pap smear
  * positive HPV test result and no control pap smear

CONTACTS AND LOCATIONS:
Overall Officials: Ken HAGUENOER, MD-PHD, Study Director — Centre de coordination des dépistages des cancers, Tours, France; Somany SENGCHANH, MD-PHD, Principal Investigator — Centre de coordination des dépistages des cancers, Tours, France
Locations (1):
- UH Tours, Tours, Indre Et Loire, France

REFERENCES:
- [Result] Boyard J, Caille A, Brunet-Houdard S, Sengchanh-Vidal S, Giraudeau B, Marret H, Rolland-Lozachmeur G, Rusch E, Gaudy-Graffin C, Haguenoer K. A Home-Mailed Versus General Practitioner-Delivered Vaginal Self-Sampling Kit for Cervical Cancer Screening: A Cluster Randomized Controlled Trial with a Cost-Effectiveness Analysis. J Womens Health (Larchmt). 2022 Oct;31(10):1472-1480. doi: 10.1089/jwh.2021.0597. Epub 2022 Jul 13. PMID 35834620